CLINICAL TRIAL: NCT03274856
Title: A Phase 2 Study to Evaluate Efficacy, Safety, and Pharmacokinetics of GLWL-01 in the Treatment of Patients With Prader-Willi Syndrome
Brief Title: A Study of GLWL-01 in Patients With Prader-Willi Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GLWL Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GLWL-PWS
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Results first posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment Sequence 1 (Other): GLWL-01 (450mg) twice a day/ Placebo
  Interventions: Drug: GLWL-01; Drug: Placebo
- Treatment Sequence 2 (Other): Placebo / GLWL-01 (450mg), twice a day
  Interventions: Drug: GLWL-01; Drug: Placebo

INTERVENTIONS:
Drug: GLWL-01 — Oral administration of 3 capsules, twice a day
Drug: Placebo — Oral administration of 3 capsules, twice a day

SUMMARY:
The aim of this study is to evaluate efficacy, safety, and pharmacokinetics of GLWL-01 in the treatment of patients with Prader-Willi Syndrome (PWS).

DETAILED DESCRIPTION:
Participants will be assigned to one of two treatment sequences (GLWL-01/Placebo or Placebo/GLWL-01), with each sequence consisting of two treatment periods separated by a washout period

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of PWS based on genetic confirmation using DNA method
* Body mass index (BMI) of 27 to 60 kg/m2
* No evidence of weight excursion beyond 10% of baseline weight
* Patients must provide assent and have a reliable caregiver (must have been caring for the patient for at least 6 months) who provides a separate written informed consent to participate. The caregiver is expected to be the primary caregiver throughout the study and must be in frequent contact with the patient (defined as at least 4 awake hours per day). The caregiver must be able to communicate with site personnel and in the investigator's opinion must have adequate literacy to complete questionnaires. If a caregiver cannot continue, 1 caregiver replacement is allowed
* Are on a stable diet and exercise regimen for >2 months prior

Exclusion Criteria:

* Current enrollment in or discontinuation within the last 30 days from a clinical trial involving any investigational drug or device
* Are currently living in a group home for more than 50% of the time
* A history or presence of other medical illness that indicates a medical problem that would preclude study participation
* Have an estimated glomerular filtration rate <60 mL/minute/1.73 m2. Have macroalbuminuria (defined as spot urine albumin to creatinine ratio of >300 μg/mg) or hematuria
* Are hypertensive (defined as sitting systolic blood pressure (BP) greater than or equal to (≥)140 millimeters of mercury (mmHg) and diastolic BP ≥90 mmHg)
* Patients on weight loss medications within 30 days of dosing, or with a history of bariatric surgery
* Unable to refrain from or anticipates the use of:

  1. Any drugs known to be significant inhibitors of Cytochrome P450, family 3, subfamily A (CYP)3A enzymes and/or P-glycoprotein (P-gp) including regular consumption of grapefruit or grapefruit juice for 14 days prior to the first dose. Acetaminophen (up to 2 grams per 24-hour period) may be permitted
  2. Any drugs known to be significant inducers of Cytochrome P450, family 3, subfamily A (CYP3A) enzymes and/or P-gp, including St. John's Wort
  3. Any medications that prolong the QT/QTc interval, unless the participant has been stable on the medication for at least 3 months and has a corrected QT interval (QTc) <450 msec
* Currently taking simvastatin >10 mg per day, atorvastatin >20 mg per day, or lovastatin >20 mg per day, or have a history of statin-induced myopathy/rhabdomyolysis
* Unsuitable for inclusion in the study in the opinion of the investigator

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — GLWL Research Inc.
Locations (7):
- United States (4):
  - Rady Children's Hospital San Diego, San Diego, California
  - University of Florida, Gainesville, Florida
  - University Hospitals, Cleveland Medical Center, Cleveland, Ohio
  - Vanderbilt University, Nashville, Tennessee
- Canada (3):
  - Alberta Diabetes Institute, University of Alberta, Edmonton, Alberta
  - CRCHUM, Montreal, Quebec
  - Centre Hospitalier Universitaire Ste-Justine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller JL, Lacroix A, Bird LM, Shoemaker AH, Haqq A, Deal CL, Clark KA, Ames MH, Suico JG, de la Pena A, Fortier C. The Efficacy, Safety, and Pharmacology of a Ghrelin O-Acyltransferase Inhibitor for the Treatment of Prader-Willi Syndrome. J Clin Endocrinol Metab. 2022 May 17;107(6):e2373-e2380. doi: 10.1210/clinem/dgac105. PMID 35213714

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Five additional participants screened but not randomized
Groups:
- Treatment Sequence 1: GLWL-01 (450mg) twice a day/ Placebo. Participants randomized to 1 of 2 treatment sequences; GLWL-01/placebo or placebo/GLWL-01 (Treatment Period 1 double-blind treatment phase/Treatment Period 2 double-blind treatment phase). During single-blind placebo lead-in phases, participants receive 3 capsules of 150-mg placebo twice daily (BID) for 14 days. During double-blind treatment phases, participants receive 3 capsules of 150-mg GLWL-01 (450 mg total dose) BID or identical placebo BID for 28 days
- Treatment Sequence 2: Placebo / GLWL-01 (450mg), twice a day. Participants randomized to 1 of 2 treatment sequences; GLWL-01/placebo or placebo/GLWL-01 (Treatment Period 1 double-blind treatment phase/Treatment Period 2 double-blind treatment phase). During single-blind placebo lead-in phases, participants receive 3 capsules of 150-mg placebo twice daily (BID) for 14 days. During double-blind treatment phases, participants receive 3 capsules of 150-mg GLWL-01 (450 mg total dose) BID or identical placebo BID for 28 days
Period: Overall Study
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2
Started | 10 | 9
Completed | 10 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Sequence 1 | Treatment Sequence 2 | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.0 (5.54) | 22.1 (4.83) | 22.1 (5.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 9 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 2 | 3 | 5
  United States | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Post-treatment Total Score on the Hyperphagia Questionnaire for Clinical Trials (HQ-CT)
Description: GLWL-01 compared with placebo on the post-treatment HQ-CT score. Total range of score of zero to 36, with higher score indicating a worse outcome.
Time Frame: Up to approximately 4 weeks of double-blind treatment
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- GLWL-01: Participants who received GLWL in either double blind treatment phase
- Placebo: Participants who received placebo in either double blind treatment phase
Arm/Group | GLWL-01 | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 15.9 (1.21) | 14.7 (1.23)

2. Secondary Outcome: Number of Participants With One or More Treatment Emergent Adverse Events (AEs) or Any Serious AEs
Description: Evaluate the safety and tolerability of GLWL-01
Time Frame: Baseline up to approximately 18 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | GLWL-01 | Placebo
Number analyzed (Participants) | 19 | 19
Participants | 8 | 7

3. Secondary Outcome: Caregiver Global Impression of Change (CGIC)
Description: GLWL-01 compared with placebo in the CGIC. Score ranges from 1 to 7, with larger number indicating a worse outcome.
Time Frame: Up to approximately 4 weeks of double-blind treatment
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | GLWL-01 | Placebo
Number analyzed (Participants) | 19 | 19
score on a scale | 4.0 (0.18) | 3.8 (0.19)

4. Secondary Outcome: Area Under the Concentration Versus Time Curve From Time Zero to 12 Hours (AUC0-12)
Description: Pharmacokinetics (PK) after single and multiple oral dosing
Time Frame: Day 14 and Day 42, pre-dose, and 0.5, 1, 2, 4, 6, and between 8 and 12 hours postdose
Population: Because PK data were collected only during Treatment 1, and the patients were randomized 1:1 to GLWL-01 or placebo, PK data were available from 9 patients. Evaluable data only available to compute AUC for some participants
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- GLWL-01 Single Dose: Day 14 observation
- GLWL-01 Multiple Dose: Day 42 observation
Arm/Group | GLWL-01 Single Dose | GLWL-01 Multiple Dose
Number analyzed (Participants) | 7 | 3
ng*h/mL | 55608 (23.6) | 121620 (23.7)

5. Secondary Outcome: Maximum Observed Drug Concentration (Cmax)
Description: Pharmacokinetics after single and multiple oral dosing
Time Frame: Day 14 and Day 42, pre-dose, and 0.5, 1, 2, 4, 6, and between 8 and 12 hours postdose
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | GLWL-01 Single Dose | GLWL-01 Multiple Dose
Number analyzed (Participants) | 9 | 9
ng/mL | 7885 (34.4) | 13695 (29.2)

ADVERSE EVENTS:
Time Frame: Up to 18 weeks
Description: Treatment-emergent adverse event: An untoward medical occurrence that emerges during a defined treatment period, having been absent pretreatment, or worsens relative to the pretreatment state, and does not necessarily have to have a causal relationship with this treatment.
Groups:
- GLWL: Participants who received GLWL in either double blind treatment phase
Arm/Group | GLWL | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 8/19 | 7/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLWL (N=19) | Placebo (N=19)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faeces soft (Gastrointestinal disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1)
Folliculitis (Infections and infestations) | 0 (0) | 1 (1)
Nail infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 3 (3) | 4 (5)
Somnolence (Nervous system disorders) | 0 (0) | 1 (2)
Agitation (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Nervous system disorders) | 0 (0) | 2 (2)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menstruation delayed (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT03274856/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/56/NCT03274856/SAP_001.pdf